CLINICAL TRIAL: NCT01919229
Title: A Randomized Pre-surgical Pharmacodynamics Study to Assess the Biological Activity of LEE011 Plus Letrozole Versus Single Agent Letrozole in Primary Breast Cancer
Brief Title: A Pharmacodynamics Pre-surgical Study of LEE011 in Early Breast Cancer Patients (MONALEESA-1)
Acronym: MONALEESA-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low recruitment, it was decided to terminate the study.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CLEE011A2201; 2013-002588-24 (EudraCT Number)
Record Dates: First submitted 2013-08-02; First posted 2013-08-08 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Early Breast Cancer
Keywords: HR-positive; HER2-negative; Breast cancer; LEE011; Letrozole; CDK; CDK4; CDK6; CDK4/6; Pharmacodynamics; Pre-surgical; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Letrozole (Active Comparator): Letrozole 2.5 mg alone once daily
  Interventions: Drug: letrozole
- LEE011 400 mg + letrozole (Experimental): Letrozole 2.5 mg once daily and ribociclib 400 mg (2 capsules of 200 mg each) once daily.
  Interventions: Drug: LEE011 (ribociclib); Drug: letrozole
- LEE011 600mg + letrozole (Experimental): Letrozole 2.5 mg once daily and ribociclib 600 mg (3 capsules of 200 mg each) once daily.
  Interventions: Drug: LEE011 (ribociclib); Drug: letrozole

INTERVENTIONS:
Drug: LEE011 (ribociclib) — Ribociclib was supplied in 200 mg hard gelatin capsules for oral use.
  Other Names: ribociclib
  Arms: LEE011 400 mg + letrozole; LEE011 600mg + letrozole
Drug: letrozole — Letrozole was supplied in 2.5mg tablets for oral use.

SUMMARY:
This is a multi-center, open-label Phase II randomized pre-surgical pharmacodynamics study.

DETAILED DESCRIPTION:
This randomized pre-surgical pharmacodynamics study will assess the biological activity of LEE011 plus letrozole versus single agent letrozole in primary breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patient is ≥ 18 years old at the time of informed consent, with newly diagnosed resectable breast cancer, who received no prior therapy for breast cancer
* Patient is postmenopausal. Postmenopausal status is defined either by:

  * Prior bilateral oophorectomy
  * Age ≥60
  * Age <60 and amenorrhea for 12 or more months and FSH (Follicle Stimulating Hormone) and estradiol in the postmenopausal range.
* Patient has a histologically (and/or cytologically) confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory.
* Patient has a grade II or grade III invasive breast cancer
* Patient has Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+ (if IHC 2+, a negative in situ hybridization (respectively FISH/CISH/SISH) test is required) by local laboratory testing
* Patient has at least one breast lesion with a diameter of ≥1.0 cm by the most accurate imaging modality used.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Patient has received any prior therapy for breast cancer.
* Patient has a concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated, basal cell skin cancer or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

  * History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to study entry
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * History of ventricular, supraventricular, nodal arrhythmias, or any other cardiac arrhythmias, Long QT Syndrome or conduction abnormality in the previous 12 months.
  * Family history of QTc prolongation or of unexplainable sudden death at <50 years of age.
  * On screening 12 lead ECG, any of the following cardiac parameters: bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval >109 msec, or QTcF >450 msec.
  * Systolic blood pressure >160 mmHg or <90 mmHg.
* Patient is currently receiving any of the following medications (see

Appendix 1 for details):

* That are known strong inducers or inhibitors of CYP3A4.
* That have a narrow therapeutic window and are predominantly metabolized through CYP3A4.
* That have a known risk to prolong the QT interval or induce Torsades de Pointes.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (4):
  - Highlands Oncology Group SC, Fayetteville, Arkansas
  - University of California at Los Angeles UCLA SC, Los Angeles, California
  - Massachusetts General Hospital SC-9, Boston, Massachusetts
  - University of Texas/MD Anderson Cancer Center Dept of MD Anderson (8), Houston, Texas
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Curigliano G, Gomez Pardo P, Meric-Bernstam F, Conte P, Lolkema MP, Beck JT, Bardia A, Martinez Garcia M, Penault-Llorca F, Dhuria S, Tang Z, Solovieff N, Miller M, Di Tomaso E, Hurvitz SA. Ribociclib plus letrozole in early breast cancer: A presurgical, window-of-opportunity study. Breast. 2016 Aug;28:191-8. doi: 10.1016/j.breast.2016.06.008. Epub 2016 Jun 20. PMID 27336726

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 patients were screened, of those 14 patients completed the Screening phase and were randomized. 6 patients discontinued during the Screening phase; 3 patients were considered screen failure and 3 patients discontinued due to patient's decision.
Groups:
- LEE011 400mg + Letrozole: Letrozole 2.5 mg once daily and ribociclib 400 mg (2 capsules of 200 mg each) once daily.
Period: Overall Study
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Started | 4 | 6 | 4
Completed | 4 | 6 | 3
Not Completed | 0 | 0 | 1
Not completed — Subject/guardian decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised of all randomized patients. Patients were analyzed according to the treatment they had been assigned to during the randomization procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole | Total
Number analyzed (Participants) | 4 | 6 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (5.48) | 64.2 (9.91) | 70.0 (4.24) | 63.8 (8.66)
Age, Customized [Number; unit: Participants]
  < 65 years | 4 | 3 | 0 | 7
  >=65 years | 0 | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 14
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cell Cycle Response Rate Per Cell Proliferation Marker Ki67
Description: Cell cycle response rate is defined by proportion of patients with natural logarithm of Ki-67 levels (expressed as percentage of baseline values) of less than 1 at the time of surgery. Since the trial was prematurely terminated, no statistical analysis was done.
Time Frame: Day 1, Day15
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Safety and Tolerability of the Combination
Description: Occurrence, frequency and severity of adverse events (AEs), laboratory abnormalities
Time Frame: Up to 30 days after the last dose
Population: Since the study was terminated, no efficacy data was obtained, but see Adverse Events (AE) section for all AEs collected.
Measure: Number; unit: Participants
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 4 | 6 | 4
Participants
  Adverse Events | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0
  Deaths | 0 | 0 | 0
  Other Adverse Events | 2 | 5 | 4

3. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Time Frame: Baseline, Day 14
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Expression of Retinoblastoma Protein (pRB)
Time Frame: Baseline, Day 15
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: PK (Pharmacokinetics) Parameters, Including But Not Limited to, Cmax, Tmax, AUClast for LEE011 (and Any Relevant Metabolites) and Letrozole.
Time Frame: Days 1, 8, 14 and 15
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in ECG Morphology
Time Frame: Baseline, Day 14
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Correlation Between PK Concentrations and ECG Changes
Description: Correlation between the QTc interval change from baseline and plasma concentrations of LEE011 and/or any relevant metabolites
Time Frame: Day 14
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Expression of Cyclin-Dependent Kinase 1 (CDK1)
Time Frame: Baseline, Day 15
Population: Since the study was terminated, no efficacy data was obtained.
Arm/Group | Letrozole | LEE011 400mg + Letrozole | LEE011 600mg + Letrozole
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Letrozole2.5mgqd: Letrozole 2.5 mg alone once daily
- LEE400mgqd+Letrozole2.5mgqd: Letrozole 2.5 mg once daily and ribociclib 400 mg (2 capsules of 200 mg each) once daily.
- LEE600mgqd+Letrozole2.5mgqd: Letrozole 2.5 mg once daily and ribociclib 600 mg (3 capsules of 200 mg each) once daily.
Arm/Group | Letrozole2.5mgqd | LEE400mgqd+Letrozole2.5mgqd | LEE600mgqd+Letrozole2.5mgqd
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 5/6 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole2.5mgqd (N=4) | LEE400mgqd+Letrozole2.5mgqd (N=6) | LEE600mgqd+Letrozole2.5mgqd (N=4)
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 3
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 2
ASTHENIA (General disorders) | 0 | 2 | 1
FATIGUE (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1
SEROMA (Injury, poisoning and procedural complications) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 2
LIPASE INCREASED (Investigations) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
BREAST PAIN (Reproductive system and breast disorders) | 1 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
HOT FLUSH (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.